CLINICAL TRIAL: NCT00353756
Title: A Placebo-Controlled, Phase 1, Single and Multiple IV Dose Escalation Study of the Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of C326 in Adults With Crohn's Disease
Brief Title: Phase 1 Study of Safety and Biological Effects of C326, an Inhibitor of IL-6, in Crohn's Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Avidia (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AV14-C001
Record Dates: First submitted 2006-07-17; First posted 2006-07-19 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-09

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

INTERVENTIONS:
Drug: C326, IL-6 Inhibitory Avimer protein

SUMMARY:
The purpose of this study is to determine whether C326, a new inhibitor of IL-6, is safe in patients with Crohn's disease.

DETAILED DESCRIPTION:
Determination of safety is the most important goal of this first study with C326. Other goals of the study are to examine:

* pharmacokinetics (change in serum concentrations over time),
* biological activity (change in blood markers relecting activity of Crohn's Disease),
* effects on symptoms of Crohn's disease.

Participants may receive either a single or several intravenous infusions of C326 or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 - 65
* Stable, moderately active Crohn's Disease
* Otherwise in generally good health

Exclusion Criteria:

* Variety of concurrent medical conditions
* Various concomitant medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52
Dates: Start 2006-09; Study Completion 2007-09

PRIMARY OUTCOMES:
Safety evaluations

SECONDARY OUTCOMES:
Pharmacokinetics
Biomarker changes -- IL-6, CRP and other acute phase reactants
Crohn's Disease Activity Index (CDAI)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Min Yap, MD, Principal Investigator — Alfred Hospital, Melbourne, Australia; Graham Radford-Smith, MD, Principal Investigator — Royal Brisbane and Womens Hospital, Brisbane, Australia
Locations (2):
- Australia (2):
  - QPharm, Brisbane, Queensland
  - Center for Clinical Studies, Melbourne, Victoria